CLINICAL TRIAL: NCT03860675
Title: Clinical Profiling, Manifestation and Assessment of Walking-related Performance Fatigability in Patients With Multiple Sclerosis: a Cross Sectional Study
Brief Title: Assessment of Walking-related Fatigability in Patients With Multiple Sclerosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FaVG-001
Record Dates: First submitted 2018-08-02; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- persons with Multiple Sclerosis (MS) (Active Comparator)
  Interventions: Diagnostic Test: Assessment of walking-related fatigability
- Healthy controls (Placebo Comparator)
  Interventions: Diagnostic Test: Assessment of walking-related fatigability

INTERVENTIONS:
Diagnostic Test: Assessment of walking-related fatigability — participants perform two six-minute walking test (6MWT), with 3-5 days in between. Before and after the 6MWT, three screenings test (spasticity, muscle strength, balance) are executed and the participants have to indicate the severity of eleven possible symptoms (= symptom inventory, SI) on a VAS scale. These screening tests and SI are continued every 10 minutes for half an hour. During a third test session, participants perform a 6-minute vigilance alphabet test in rest and while doing a 6MWT to investigate the relationship between cognitive and motor fatigability.

SUMMARY:
The primary goal of this interventional study is to objectively examine the prevalence of walking-related performance fatigability, together with the psychometric properties of its measuring parameters. The secondary aim is to investigate the relation of other clinical symptoms to walking-related performance fatigability.

The following three research questions will be addressed:

1. How prevalent is walking-related performance fatigability and what are the psychometric properties of fatigability formulas in preparation of use as experimental outcome measure?
2. What are associated symptoms of walking-related motor fatigability and how long does this manifest?
3. What is the relationship between cognitive fatigability and walking-related performance fatigability?

participants perform two six-minute walking test (6MWT), with 3-5 days in between. Before and after the 6MWT, three screenings test (spasticity, muscle strength, balance) are executed and the participants have to indicate the severity of eleven possible symptoms (= symptom inventory, SI) on a VAS scale. These screening tests and SI are continued every 10 minutes for half an hour. During a third test session, participants perform a 6-minute vigilance alphabet test in rest and while doing a 6MWT to investigate the relationship between cognitive and motor fatigability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 70 years
* Confirmed diagnosis according to the McDonald criteria
* Performed a 6MWT before, to ensure familiarization
* Able to walk independently or with unilateral support for 6 minutes without rest
* Signed the informed consent

Exclusion Criteria:

* Exacerbation or relapse within last 3 months before study
* Other neurological diagnosis, such as stroke and Parkinson
* MS-like syndromes, such as neuromyelitis optica
* Other medical condition interfering with walking ability (e.g. cardiac or respiratory diseases, arthritis and fibromyalgia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Deceleration index | day 1
  Formula for walking-related performance fatigability: (distance min6 - distance min1)/(distance min1) x100 Cut-off value: -15%

SECONDARY OUTCOMES:
Symptom Inventory Questionnaire | day 1
  Visual analog scale for the 11 symptoms of the SI: General fatigue, motor fatigability, attention problems, spasticity, sensitivity, visual disturbance, balance disturbance, gait pattern impairments, pain, dizziness, muscle weakness (pre/post/10'post/20'post/30'post 6MWT)
Symptom Inventory Questionnaire | day 4
  Visual analog scale for the 11 symptoms of the SI: General fatigue, motor fatigability, attention problems, spasticity, sensitivity, visual disturbance, balance disturbance, gait pattern impairments, pain, dizziness, muscle weakness (pre/post/10'post/20'post/30'post 6MWT)
spasticity | day 1
  Modified Ashworth Scale for spasticity (0 - 1 - 1+ - 2 - 3 - 4) (pre/post/10'post/20'post/30'post 6MWT)
spasticity | day 4
  Modified Ashworth Scale for spasticity (0 - 1 - 1+ - 2 - 3 - 4) (pre/post/10'post/20'post/30'post 6MWT)
Strength | day 1
  Motricity Index for muscle strength (0 - 9 - 14 - 19 - 25 - 33) (pre/post/10'post/20'post/30'post 6MWT)
Strength | day 4
  Motricity Index for muscle strength (0 - 9 - 14 - 19 - 25 - 33) (pre/post/10'post/20'post/30'post 6MWT)
Balance | day 1
  Romberg test for balance (pre/post/10'post/20'post/30'post 6MWT)
Balance | day 4
  Romberg test for balance (pre/post/10'post/20'post/30'post 6MWT)
VAS fatigue | day 1
  Visual analog scale for fatigue pre 6MWT and after each minute of 6MWT (0 - 1 - 2 - 3 - 4 - 5 - 6 - 7 - 8 - 9 - 10)
VAS fatigue | day 4
  Visual analog scale for fatigue pre 6MWT and after each minute of 6MWT (0 - 1 - 2 - 3 - 4 - 5 - 6 - 7 - 8 - 9 - 10)
heart rate | day 1
  Heart rate pre 6MWT and after each minute of 6MWT
heart rate | day 4
  Heart rate pre 6MWT and after each minute of 6MWT
gait parameter | day 1
  APDM opal sensors: sensors to analyze the spatiotemporal parameters of gait while walking for 6minutes.
gait parameter | day 4
  APDM opal sensors: sensors to analyze the spatiotemporal parameters of gait while walking for 6minutes.
Cognitive fatigability | between week 1 and week 2 (no specific day: at the day the patients request)
  deceleration of reaction time of answers of the Alphabeth vigilance test six minutes while walking and the Alphabeth vigilance test six minutes in rest.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Fanny Van Geel, drs., Study Chair — Hasselt University
Locations (3):
- Belgium (3):
  - Hasselt University, Diepenbeek
  - National MS Center Melsbroek, Melsbroek
  - Revalidatie & MS Centrum Overpelt, Overpelt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Van Geel F, Bielen H, Theunissen K, Moumdjian L, Van Nieuwenhoven J, Van Wijmeersch B, Meesen R, Ramari C, Feys P. Clinical manifestation and perceived symptoms of walking-related performance fatigability in persons with multiple sclerosis. Int J Rehabil Res. 2021 Jun 1;44(2):118-125. doi: 10.1097/MRR.0000000000000457. PMID 33534273
- [Derived] Van Geel F, Veldkamp R, Severijns D, Dalgas U, Feys P. Day-to-day reliability, agreement and discriminative validity of measuring walking-related performance fatigability in persons with multiple sclerosis. Mult Scler. 2020 Nov;26(13):1785-1789. doi: 10.1177/1352458519872465. Epub 2019 Sep 9. PMID 31496362